

## Protocol for non-interventional studies based on existing data

| Document Number: | c30353958-01 |
|---|---|
| BI Study Number: | 0135-0344 |
| BI Investigational Product(s): | Actilyse |
| Title: | Safe Implementation of Treatments in Stroke (SITS) - |
| | Intravenous thrombolysis in acute ischaemic stroke patients over 80 years, SITS-IVT>80 years study |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | na |
| PASS: | Yes |
| EU PAS register number: | Study not yet registered |
| Active substance: | Alteplase |
| Medicinal product: | Actilyse: Powder and solvent for solution for injection |
| | and infusion, 10 mg, 20 mg, and 50 mg |
| <b>Product reference:</b> | DE/H/0015/004 |
| Procedure number: | DE/H/0015/004/IB/135 |
| Joint PASS: | No |
| Research question and objectives: | Pooled analysis of randomized controlled trials (RCTs) of intravenous thrombolysis (IVT) with Alteplase, a recombinant tissue plasminogen Activator (rt-PA) for acute ischemic stroke, has shown that patients >80 years treated with IVT versus control derived equal benefit compared to patients 18-80 years. The SITS-ISTR (Safe Implementation of Treatment in Stroke-International Stroke Thrombolysis Register)-VISTA analysis demonstrated benefit of IVT in patients >80 years compared to control, and found no difference in the slope of benefit versus treatment delay for younger versus elderly patients <sup>3</sup> , a finding that was confirmed in the RCT dataset. The European guideline recommends use of IVT within 4.5h of symptom onset also in the elderly. Until recently, most European regulatory agencies |

| | had not approved marketing of IVT with Alteplase for use in ischemic patients >80 years. A recently published SITS study showed that unselected patients >80-years treated with IVT after 3h versus earlier, had a slightly higher rate of SICH but similar unadjusted functional outcome and poorer adjusted outcome. IVT with Alteplase in >80 years old patients treated within 4.5h of symptom onset is now approved in a number of European and non-European countries. Safety and outcome of a treatment in acute ischaemic stroke may be different in the RCT settings in patients over 80 years. Although IVT in patients >80 years has been used off-label in many countries prior to approval, use of IVT in patients>80 years will probably be more frequent after approval. The proposed SITS-ISTR provides an opportunity for continuous monitoring of thrombolysis treatment in stroke, and provides a |
|---|---|
| | technical foundation for the SITS->80 years post-approval study. The SITS-IVT>80 years is a retrospective study based on data collected in the SITS-ISTR setting from acute ischemic stroke patients > 80 years of age. The study aims to evaluate the incidence rate with 95% CI of SICH, death and functional independence/favourable outcome within 90 days for ischaemic stroke patients treated with rt-PA in clinical routine settings. In the proposed SITS-IVT>80 years study using the SITS registry we plan to identify approximately 1000 patients older than 80 years treated with IV Alteplase otherwise fulfilling SmPC criteria in the post-approval period of 3 years (from 1 July 2018 to 30 June 2021) and also to identify 1000 patients older than 80 years treated with IV Alteplase otherwise fulfilling SmPC criteria in the pre-approval period of 3 years (from June 2015 to June 2018). In both periods, at least 500 patients should be registered from centres of European countries being part of the mutual recognition. The objective of the SITS-IVT>80 years is to compare the safety and other outcome parameters between the post-approval >80 |
| | years and pre-approval >80 years AIS patients using the data already collected in SITS-ISTR. |
| Country(-ies) of study: | Austria, Belgium, Cyprus, Germany, Denmark, Greece, Spain, Finland, France, Ireland, Iceland, Italy, Luxemburg, Malta, Netherland, Norway, Portugal, Sweden, United Kingdom |
| Author: | Phone |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Marketing authorisation holder(s): | |
|---|---|
| MAH contact person: | |
| EU-QPPV: | Boehringer Ingelheim International GmbH Binger Strasse 173 55216 Ingelheim am Rhein |
| Signature of EU-QPPV: | |
| Date: | 25 Nov 2019 |
| Proprietary confidential information<br>© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved | |

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

01- MCS-90-124\_RD-01 (4.0)

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 1. TABLE OF CONTENTS

| TITLE PAGE | 1 |
|------------------------------------------|----|
| 1. TABLE OF CONTENTS | 4 |
| 2. LIST OF ABBREVIATIONS | 6 |
| 3. RESPONSIBLE PARTIES | 8 |
| 4. ABSTRACT | 10 |
| 5. AMENDMENTS AND UPDATES | 15 |
| 6. MILESTONES | 16 |
| 7. RATIONALE AND BACKGROUND | 17 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 20 |
| 9. RESEARCH METHODS | 21 |
| 9.1 STUDY DESIGN | 21 |
| 9.2 SETTING | 21 |
| 9.2.1 Level of care | 21 |
| 9.3 VARIABLES | 22 |
| 9.3.1 Exposures | 22 |
| 9.3.2 Outcomes | 23 |
| 9.3.2.1 Primary outcomes | 23 |
| 9.3.2.2 Secondary outcomes | 23 |
| 9.3.3 Covariates | 24 |
| 9.4 Onset to treatment time DATA SOURCES | 25 |
| 9.5 STUDY SIZE | 25 |
| 9.6 DATA MANAGEMENT | 25 |
| 9.7 DATA ANALYSIS | 25 |
| 9.7.1 Main analysis | 26 |
| 9.8 QUALITY CONTROL | |
| 9.8.1 Investigators and local procedures | 27 |
| 9.9 LIMITATIONS OF THE RESEARCH METHODS | 28 |
| 9.10 OTHER ASPECTS | 28 |
| 9.11 SUBJECTS | 29 |

| Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of | its affiliated companies |
|---|---|
| 9.11.1 Cases | 29 |
| 9.11.2 Controls | 29 |
| 9.12 BIAS | 29 |
| 10. PROTECTION OF HUMAN SUBJECTS | 30 |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 31 |
| 12. AS AN OBSERVATIONAL STUDY, BASED ON EXIDATA, ALL PATIENT DATA IS DE-IDENTIFIED AN BE ANALYSED IN AGGREGATE. INDIVIDUAL PA SAFETY RELATED INFORMATION WILL NOT BE CAPTURED DURING THIS STUDY. THUS, INDIVIDUAL SAFETY REPORTING IS NOT APPLICABLE. SAFET REPORTING WILL BE DONE CUMULATIVELY IN AGGREGATE IN THE STUDY REPORT.PLANS FOR DISSEMINATING AND COMMUNICATING STUDY | ND WILL TIENT DUAL TY |
| RESULTS | 31 |
| 13. REFERENCES | 32 |
| 13.1 PUBLISHED REFERENCES | 32 |
| ANNEX 1. LIST OF STAND-ALONE DOCUMENTS | 36 |
| ANNEX 2. ENCEPP CECKLIST FOR STUDY PROTOCOL | LS37 |
| ANNEX 3. ADDITIONAL INFORMATION | 44 |

**Study Number 0135-0344** 

c30353958-01

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

AE Adverse Event

AUC Area under the Curve
CI Confidence Interval
CML Local Clinical Monitor
CRA Clinical Research Associate

CRF Case Report Form CT Computer Tomogram

CTCAE Common Terminology Criteria for Adverse Events

CTMF Clinical Trial Master File
CTP Clinical Trial Protocol
CTR Clinical Trial Report

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

EU European Union

EudraCT European Clinical Trials Database

FAS Full Analysis Set
GCP Good Clinical Practice
HPC Human Pharmacology Centre

IB Investigator's Brochure

ICO International Coordinating OfficeIEC Independent Ethics CommitteeIRB Institutional Review BoardISF Investigator Site File

i.v. intravenous

IVRS Interactive Voice Response System
IWRS Interactive Web-based Response System

MedDRA Medical Dictionary for Drug Regulatory Activities

MCA Middle Cerebral Artery
MRI Magnetic Resonance Imaging

MST Medical Subteam

NIHSS National Institute of Health's Stroke Scale

OPU Operative Unit p.o. per os (oral)

PCC Protocol Challenge Committee
PH Parenchymal Haemorrhage
q.d. quaque die (once a day)
SAE Serious Adverse Event

s.c. Subcutaneous

SICH Symptomatic Intracerebral Haemorrhage SmPC Summary of Product Characteristics SPC Summary of Product Characteristics

SITS-ISTR Safe Implementation of Treatments in Stroke- International Stroke

Thrombolysis Registry

TCM Trial Clinical Monitor

### **Boehringer Ingelheim**

**Study Number 0135-0344** 

### Protocol for non-interventional studies based on existing data

c30353958-01

**** 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TDMAP Trial Data Management and Analysis Plan

t.i.d. ter in die (3 times a day)

t-PA Tissue plasminogen activator, alteplase, Actilyse®

TMM Team Member Medicine TMW Trial Medical Writer

TSAP Trial Statistical Analysis Plan

**Study Number 0135-0344** 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. **RESPONSIBLE PARTIES**

#### SITS ORGANISATION

SITS International: Responsibility: Representatives: SITS Scientific Committee • Scientific responsibility • Data evaluation • Monitoring SITS Scientific activities, e.g. projects, reports and publications Data management Data management and statistical analysis Statistical support will also be sought from Manage centre application, SITS ICO (International coordinate, maintain and Coordination Office) online monitoring of SITS registry, development and maintenance of database





On behalf of Boehringer Ingelheim International GmbH:

### Boehringer Ingelheim Protocol for non-interventional studies based on existing data Study Number 0135-0344

**** 

c30353958-01

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Boehringer Ingelheim Binger Strasse 173 55216 Ingelheim am Rhein Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 4. ABSTRACT

| Name of con | npany: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| <b>product:</b> If applicable, | shed medicinal list centrally- edicinal product(s) estudy. | | |
| List pharmac group(s){AC | ive ingredient: otherapeutic T codes} and active subject to the study | | |
| Protocol | Study number: | Version/Revision: | Version/Revision date: |
| date:<br>25 Nov<br>2019 | 0135-0344 | 1.0 | |
| Title of study: | A non-interventional rt-PA (0.9 mg/kg) in to the Summary of P | ion of Treatments in Stroke (SITS) - Intravenous thrombolysis in croke patients over 80 years, SITS-IVT>80 years study. nal post-approval study on SITS-ISTR existing data of intravenous in acute ischaemic stroke patients over 80 years, treated according f Product Characteristics (SmPC) of European countries being part ognition procedure within the academic SITS-ISTR (International | |
| Rationale<br>and<br>backgroun<br>d: | Pooled analysis of randomized controlled trials (RCTs) of intravenous thrombolysis (IVT) with Alteplase, a recombinant tissue plasminogen Activator (rt-PA) for acute ischemic stroke, has shown that patients >80 years treated with IVT versus control derived equal benefit compared to patients 18-80 years. Effectiveness of IVT diminished as the treatment delay increased across the first 6 hours without a corresponding increase in the relative risk of symptomatic intracerebral hemorrhage (SICH). Real world registry experience supports these RCT data in patients >80 years treated within 3h. The SITS-ISTR (Safe Implementation of Treatment in Stroke-International Stroke Thrombolysis Register)-VISTA analysis demonstrated benefit of IVT in patients >80 years compared to control, and found no difference in the slope of benefit versus treatment delay for younger versus elderly patients, a finding that was confirmed in the RCT dataset. Until recently, most European regulatory agencies had not approved marketing of IVT with Alteplase for use in ischemic patients >80 years, whereas the American regulatory agency supports promotion of IVT in patients >80 years within 3h of symptom onset. A recently published SITS study showed that unselected patients >80-years treated with IVT after 3h versus earlier, had a slightly higher rate of SICH but similar unadjusted functional outcome and poorer adjusted outcome. The European guideline | | |

| Name of con | nnanv: | | |
|---|---|---|---|
| Boehringer In | | | |
| Name of fini product: If applicable, | ished medicinal list centrally- edicinal product(s) | | |
| Name of acti<br>List pharmac<br>group(s){AC | ive ingredient: | | |
| Protocol | Study number: | Version/Revision: | Version/Revision date: |
| date:<br>25 Nov<br>2019 | 0135-0344 | 1.0 | |
| Research | Safety and outcome RCT settings in paticused off-label in markill probably be more opportunity for conting provides a technical SITS-IVT>80 years acute ischaemic paticular characteristics (Smisich, death and ind stroke patients over 2000 patients overal identified for the SIT will be compared be patients. | e of a treatment in acute ischaemic stroke may be different in the tients over 80 years. Although IVT in patients >80 years has been any countries prior to approval, use of IVT in patients>80 years for frequent after approval. The SITS-ISTR setting provides an antinuous monitoring of thrombolysis treatment in stroke, and all foundation for the SITS->80 years post-approval registry. The is a retrospective study of existing data in the SITS-ISTR on attents treated with IVT according to the Summary of Product anPC) criteria. The study aims to evaluate the incidence rate of adependence/favourable outcome within 90 days for ischaemic ar 80 years treated with rt-PA in clinical routine settings. At least all from approximately 60 European sites are planned to be ITS-IVT>80 years study. Safety and other outcome parameters between post-approval >80 years and pre-approval >80 years | |
| Research<br>question<br>and<br>objectives: | Safety and outcome of a treatment in acute ischaemic stroke may be different in the RCT settings in patients over 80 years. Although IVT in patients >80 years has been used off-label in many countries prior to approval, use of IVT in patients>80 years will probably be more frequent after approval. The study aims to evaluate the incidence rate of SICH, death and independence/favourable outcome within 90 days for ischaemic stroke patients treated with rt-PA in clinical routine settings. The SITS-IVT>80 years Study will primarily investigate the safety and outcome of IVT in acute ischaemic stroke in patients >80 years collected during the post-approval period and to compare the safety outcome with existing pre-approval patients >80 years collected in routine clinical practice and recorded in the SITS registry. | | |

| Name of con | npany: | | |
|---|---|---|---|
| Boehringer In | ngelheim | | |
| Name of finished medicinal product: If applicable, list centrally-authorised medicinal product(s) subject to the study. | | | |
| List pharmac<br>group(s){AC<br>substance(s) | ive ingredient: otherapeutic T codes} and active subject to the study | | |
| Alteplase | T | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 25 Nov<br>2019 | 0135-0344 | 1.0 | |
| Study design: | This is a retrospective | ve observational study using existing | ng data from the SITS registry. |
| Population: | Post-approval: Patients over 80 years old presenting with acute ischaemic stroke symptoms for which thrombolysis treatment was initiated within 4.5 hours after stroke onset according to the SmPC during the study period July 2018 to June 2021. Pre-approval: Patients aged over 80 years presenting with acute ischaemic stroke symptoms for which thrombolysis treatment was initiated within 4.5 hours after stroke onset otherwise according to SmPC during the period of approximately 3 years prior to approval (June 2015 to June 2018) | | |
| Variables: | Standard SITS-ISTR | R safety parameters: | |
| | <ul> <li>Symptomatic intracerebral haemorrhage (SICH):</li> <li>Intracerebral haemorrhage (parenchymatous haemorrhage type 2), at post-treatment scan combined with neurological deterioration leading to an increase of 4 points on the NIH Stroke Scale (SITS-MOST definition)</li> <li>Mortality:</li> <li>Death (mRS = 6) at day 90</li> </ul> | | |
| | Independence / favourable outcome: | | |
| | Independence for the activities of daily living at day 90. Good functional outcome is defined as a modified Rankin Scale (mRS) score of both 0-2 (independence) and 0-1 (favourable) | | |
| | | and demographic variables available in the SITS registry for g patient characteristics. | |
| | | anagement variables | |
| | o Time from onset to door | | |
| | Door to needle (treatment) time | | |

| Name of con | npany: | | |
|---|---|---|---|
| Boehringer In | ngelheim | | |
| Name of finished medicinal product: If applicable, list centrally-authorised medicinal product(s) subject to the study. | | | |
| List pharmac group(s){AC | otherapeutic T codes} and active subject to the study | | |
| Protocol | Study number: | Version/Revision: | Version/Revision date: |
| date:<br>25 Nov<br>2019 | 0135-0344 | 1.0 | |
| | o Ons | et to treatment time | |
| Data sources: | The SITS-ISTR | | |
| Study size: | SmPC after approva<br>treated with IV Alte<br>approval of the indic<br>and post-approval po-<br>registry. The sample | 000 patients above 80 years treated with IV Alteplase according to oval of indication and approximately 1000 patients above 80 years Alteplase within 4.5 hours otherwise according to SmPC before the indication. Of these at least 500 patients each from the pre-approval all period from centres of European countries being part of SITS inple size of the study is not based on any formal power calculation, insultation with authorities, based on numbers considered to be in a 3-year period. | |
| Data<br>analysis: | groups. Multivariabl | loratory analyses in the unmatched le analysis with adjustment for diff for outcome comparisons. | |
| Milestones: | Post approval data collection is Q3 2018 or Q2 | | imated timelines<br>3 2018 or Q2 2021<br>ast patient out October 2021 |
| | Interim rep | orts Ye | early |
| | | t to be available within 6 Apole he database lock | pril 2022 |
| | _ | t to be submitted two Ju<br>er its availability | ne 2022 |

### Boehringer Ingelheim Protocol for non-interventional studies based on existing data Study Number 0135-0344


c30353958-01

| Name of con | ipany: | | |
|---|---|---|---|
| Boehringer In | ngelheim | | |
| <b>product:</b> If applicable, | list centrally-edicinal product(s) | | |
| List pharmac<br>group(s){AC<br>substance(s) | otherapeutic T codes} and active subject to the study | | |
| Alteplase | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 25 Nov<br>2019 | 0135-0344 | 1.0 | |
| | Re-assessment of the | e timelines will be performed as stud | dy progresses |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. AMENDMENTS AND UPDATES

None

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. MILESTONES

| Planned milestones | Estimated timelines |
|---|---|
| Post approval data collection is planned after the majority of the participating countries received approval of the label change for >80 years with acute ischaemic stroke | Q3 2018 or Q2 2021<br>Last patient out October 2021 |
| Interim reports | Yearly |
| Final report to be available within 6 months of the database lock | April 2022 |
| Final report to be submitted two months after its availability | June 2022 |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RATIONALE AND BACKGROUND

#### Stroke – a growing disease

Stroke is the third leading cause of death and the number one cause of neurological disability in adults globally, not only in the elderly, but also in younger age groups. Labout one million strokes occur annually within the European Union. Stroke patients often require extended hospital stays followed by rehabilitation, ongoing support from the community, and nursing-home care.

Alarmingly, stroke incidence is expected to increase considerably over the next decades because of an increase in the elderly population. The proportion of people over the age of 70, which was 13% in year 2000, is expected to be 20% in year 2050. It is predicted that stroke will account for 6.2% of the total burden of illness in 2020. Thus, without major advances to improve prevention and treatment, the cost of this disease will increase dramatically. 3.4

#### Treatment strategies for stroke

Stroke unit care  $^{5.6}$  and reperfusion therapy by iv thrombolysis within 4.5 hours of symptom onset  $^{7-12}$ , and/or endovascular thrombectomy within 6 hours of symptom onset in anterior circulation stroke  $^{13-19}$ , are the only evidence-based treatments for acute ischemic stroke, and are recommended by national and international practice guidelines.  $^{20-21}$ 

#### Stroke unit care

Stroke unit care is the evidence-based treatment for patients with all types of acute stroke in all ages and severity grades. The aggregate of multidisciplinary treatment, monitoring and care measures in dedicated stroke units prevents complications, improves functional outcomes, and reduces stroke mortality. Stroke unit care increases chance of independent survival by an absolute of 5-6 % compared to treatment in general medical wards, and the effect is sustainable for 10 years or more. <sup>5,6</sup> In Sweden, approximately 91 % of all stroke patients are admitted to a stroke unit. <sup>1</sup>

#### Intravenous thrombolysis

Intravenous thrombolysis with tissue plasminogen activator (tPA) within 4.5 hours of ischaemic stroke onset is an established and approved treatment<sup>7-12</sup>. The effect of iv thrombolysis is time-dependent. Among patients treated within one hour, every second patient is expected to fully recover within three months, among those treated within 90 minutes, every third, and within 3 hours every seventh patient. For patients treated within the time interval of 3-4.5 hours, 14 patients need to be treated for one additional patient to recover fully. IV thrombolysis given within three hours from stroke onset increases the chance of reaching good functional outcome (defined as having exactly the same functional level as before the stroke) from 23% to 33%, and when given between 3 and 4.5 hours from onset, by a more modest but still substantial absolute 5%. The use of iv thrombolysis is increasing but still used in only 10-15% of all ischaemic stroke patients. Meanwhile, 2-7% of patients treated with iv thrombolysis suffer symptomatic intracerebral haemorrhage (ICH) as a complication, leading to death in 1.5-2%, and worsening functional outcome in survivors. <sup>8,9</sup>


c30353958-01

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Endovascular thrombectomy Endovascular thrombectomy, 13-19 although highly effective in reducing stroke disability and potentially mortality, is only indicated in large artery occlusion, feasible in a minority of patients, and is most commonly used in addition to iv thrombolysis.

#### The rationale for thrombolytic treatment

Thromboembolic occlusion of an artery leading to the brain or in the brain, is a major cause of stroke. An occlusion of an artery leads to immediate drop of blood flow into the corresponding arterial territory. The size and site of the occlusion, and the efficiency of compensatory flow through collateral arteries determine the amplitude and the extension of the drop in the blood flow. If the flow is reduced to about 20 ml/100 g/minute (about 40% of the normal value), neurological symptoms occur. A blood flow below 10 ml/100 g/min is not compatible with cell survival, and the brain tissue is infarcted. Brain tissue with a blood flow between 10 and 20 ml/100g/min may survive for a few hours, but is likely to die if blood flow is not re-established.<sup>2</sup>

Spontaneous reperfusion may occur through endogenous release of plasminogen activator, which stimulates plasmin formation from plasminogen. For larger occlusions, this release seems insufficient to induce reperfusion in time to avoid a cerebral lesion.

Administration of plasminogen activator as an intravenous infusion is thus a method to enhance this endogenous procedure. Reperfusion should of course be done as early as possible to avoid a cerebral lesion, and to avoid complications caused by ischaemic injury to blood vessel walls and the blood-brain barrier.

#### Evidence from randomised controlled trials

In total, 17 randomised trials with 5,216 patients form the evidence base for thrombolysis in stroke. Of the data derived from these trials, 42% relate to streptokinase, 3% to intravenous urokinase and 5% to intra-arterial pro-urokinase. 50% of the data comes from trials using intravenous rt-PA. The results of these trials and agents are frequently discussed together, which may give a more unfavourable impression of the effect of thrombolysis than if only intravenous rt-PA is studied. Whether there is true heterogeneity between thrombolytic agents is still not quite clarified, but there are differences between e.g. streptokinase and rt-PA in the effect on blood pressure (streptokinase reduces blood pressure) which may cause differential effects on collateral blood flow to the ischaemic area of the brain.

A meta-analysis<sup>9</sup> of individual patient data from 6756 patients in 9 randomised trials 7,11,23-27 comparing intravenous thrombolysis with Alteplase with placebo or open control in acute ischemic stroke shows that Alteplase significantly improves the overall odds of a good stroke outcome (defined by a modified Rankin score (mRS) of 0-1) when given within 4.5 h of stroke onset. The earlier treatment is associated with higher proportional benefits. Although Alteplase treatment significantly increased the odds of symptomatic intracranial haemorrhage and of fatal intracranial haemorrhage within 7 days but by 3-6 months this risk was offset by an average absolute increase in disability- free survival of about 10% for patients treated within 3 hours and about 5% for patients treated between >3 and 4.5 hours.

For rt-PA, data from 2,955 patients are available for analysis. Of these, 869 were included within three hours after onset of clinical symptoms. The results are more favourable for patients included within three hours compared to those included between three and six hours. The number needed to treat to get one more favourable outcome increases from 4.5, during the first 90 minutes, to 9 between 1.5 and 3 hours, and to 14 between 3 and 4.5 hours.  $\frac{28}{100}$ 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Pooled analysis of randomized controlled trials (RCTs) of intravenous thrombolysis (IVT) with Alteplase, a recombinant tissue plasminogen Activator (rt-PA) for acute ischemic stroke, has shown that patients >80 years treated with IVT versus control derived equal benefit compared to patients 18-80 years. Effectiveness of IVT diminished as the treatment delay increased across the first 6 hours without a corresponding increase in the relative risk of symptomatic intracerebral haemorrhage (SICH). Real world registry experience supports these RCT data in patients >80 years treated within 3h. The SITS-ISTR (Safe Implementation of Treatment in Stroke-International Stroke Thrombolysis Register)-VISTA analysis demonstrated benefit of IVT in patients >80 years compared to control, and found no difference in the slope of benefit versus treatment delay for younger versus elderly patients, a finding that was confirmed in the RCT dataset.

### Experiences from post-trial treatments

Several open studies have been performed to address the issue of safety and efficacy of routine thrombolysis in acute stroke<sup>29-34</sup>. In the absence of control groups, the outcome of these studies must be compared with the results of randomised controlled trials. Such comparisons have been difficult since the baseline characteristics in most of the studies have not been comparable. This is illustrated by Katzan et al<sup>31</sup> who reported the highest rate of cerebral haemorrhages of all studies. Initial stroke severity, the most important predictor of haemorrhagic complication risk was reported in only 40 % of all patients and in only 27 % of those with haemorrhage.

#### Guideline recommendation and approval status

The European guideline<sup>38</sup> recommends use of IVT within 4.5h of symptom onset also in the elderly, but North American guidance does not recommend IVT in the >3-4.5h window in patients >80 years.<sup>39</sup> Until recently, most European regulatory agencies had not approved marketing of IVT with Alteplase for use in ischemic patients >80 years, whereas the American regulatory agency supports promotion of IVT in patients >80 years within 3h of symptom onset. A recently published SITS study showed that unselected patients >80-years treated with IVT after 3h versus earlier, had a slightly higher rate of SICH but similar unadjusted functional outcome and poorer adjusted outcome.<sup>40</sup> IVT with Alteplase within 4.5h of symptom onset is now approved in a number of European and non-European countries.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8. RESEARCH QUESTION AND OBJECTIVES

Safety and efficacy of a treatment in acute ischaemic stroke may be different in the RCT settings in patients over 80 years. Although IVT in patients >80 years has been used off-label in many countries prior to approval, use of IVT in patients>80 years will probably be more frequent after approval. The SITS-ISTR provides an opportunity for continuous monitoring of thrombolysis treatment in stroke, and provides a technical foundation for the SITS->80 years post-approval registry. The proposed SITS-IVT>80 years is a retrospective study of existing data in the SITS-ISTR for the ischaemic stroke patients treated with IVT according to the Summary of Product Characteristics (SmPC) criteria. The study aims to evaluate the incidence rate of SICH, death and independence/favourable outcome within 90 days for ischaemic stroke patients treated with rt-PA in clinical routine settings. At least 2000 (1000 in the post-approval and 1000 in the pre-approval) patients overall from approximately 60 European sites are planned to be identified in the SITS-IVT>80 years study. Safety and other outcome parameters will be compared between post-approval >80 years and pre-approval >80 years patients.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

The SITS-IVT>80 years is an observational, multinational, multicenter study in patients with acute ischaemic stroke treated with IV thrombolysis according to SmPC. This is a retrospective study based on existing data collected in the registry for patients treated according to the revised and approved Summary of Product Characteristics (SmPC) of IVT>80 years in European countries.

Approximately 1000 patients older than 80 years treated with IV Alteplase are expected to be identified for the proposed SITS-IVT>80 year study in the post-approval period of 3 years (1 July 2018 to 30 June 2021) and also approximately 1000 patients above 80 years treated with IV Alteplase within 4.5 hours otherwise according to SmPC in the pre-approval period (June 2015 to June 2018). Of these, at least 500 patients each should be registered from European centers (see list of European countries being part of the mutual recognition procedure) during the pre-approval as well as in the post-approval period. If the target 1000 patient is not reached during the 3 year period (post-approval phase), the data exchange will stop provided at least 500 patients registered from European centers have been included into the analysis.

The aim is to investigate the incidence rate of SICH, death and functional independence (mRS) / favorable outcome (primary endpoints) at day 90 in post-approval registered group of >80 year old patients and to compare with pre-approval registered group of >80 year old patients, comparison will be in both unmatched and the propensity score matched groups in the SITS-ISTR registry.

Additional analyses will be made with regards to patient's characteristics, management time (secondary endpoints): onset of symptoms to time of treatment initiation, and its components: onset of symptoms to door; door to treatment initiation.

#### 9.2 SETTING

The SITS-IVT>80 years Study is driven by the SITS International according to SITS policy, and data will be provided to the Regulatory Authorities as needed. Acute ischaemic stroke patients aged >80 years who received IV thrombolysis according to SmPC during the period June 2015 to June 2021 were considered. Of these, pre-approval sample will consist at least 1000 patients from June 2015 to June 2018 and post-approval sample of 1000 patients from July 2018 to June 2021.

#### 9.2.1 Level of care

• Thrombolysis treatment should be given at a semi-intensive care unit within a stroke unit, or an intensive care unit or semi-intensive care unit in close collaboration with the stroke unit, under the responsibility of an experienced stroke neurologist/stroke

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

physician. This stroke neurologist/stroke physician should have personal experience from thrombolysis treatment in stroke.

#### Inclusion criteria

- Patients over 80 years old presenting with acute ischaemic stroke symptoms for which thrombolysis treatment was initiated within 4.5 hours after stroke onset according to SmPC are included.
- Patients over 80 years who received thrombolysis according to SmPC for AIS within 4.5 hours after stroke onset during the period (approximately 3 years) prior to July 2018 are included.

#### Exclusion criteria

- Contraindication(s) to the use of IV thrombolysis per local SmPC.
- Documentation that the patient was enrolled or is planned to be enrolled in an investigational clinical trial at the time of the onset of index event and for the duration of the data collection.

#### 9.3 VARIABLES

### 9.3.1 Exposures

#### <u>Intravenous thrombolysis</u>

Index date is defined as the date of initiation of IV thrombolysis with alteplase (Actilyse<sup>®</sup>).

Intravenous thrombolysis with tissue plasminogen activator (tPA) within 4.5 hours of ischaemic stroke onset is an established and approved treatment. The effect of iv thrombolysis is time-dependent. Among patients treated within one hour, every second patient is expected to fully recover within three months, among those treated within 90 minutes, every third, and within 3 hours every seventh patient. For patients treated within the time interval of 3-4.5 hours, 14 patients need to be treated for one additional patient to recover fully. IV thrombolysis given within three hours from stroke onset increases the chance of reaching good functional outcome (defined as having exactly the same functional level as before the stroke) from 23% to 33%, and when given between 3 and 4.5 hours from onset, by a more modest but still substantial absolute 5%. The use of iv thrombolysis is increasing but still used in only 10-15% of all ischaemic stroke patients. Meanwhile, 2-7% of patients treated with iv thrombolysis suffer symptomatic intracerebral haemorrhage (ICH) as a complication, leading to death in 1.5-2%, and worsening functional outcome in survivors. So

Administration of plasminogen activator as an intravenous infusion is thus a method to enhance this endogenous procedure. Reperfusion should of course be done as early as possible to avoid a cerebral lesion, and to avoid complications caused by ischaemic injury to blood vessel walls and the blood-brain barrier.

Treatment with Actilyse must be started as early as possible within 4.5 hours of the onset of symptoms. Beyond 4.5 hours after onset of stroke symptoms there is a negative benefit risk ratio associated with Actilyse administration and so it should not be administered.

**Study Number 0135-0344** 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The recommended total dose is 0.9 mg alteplase/kg body weight (maximum of 90 mg) starting with 10% of the total dose as an initial intravenous bolus, immediately followed by the remainder of the total dose infused intravenously over 60 minutes.

Patients in general will be exposed once to Actilyse for the treatment of the acute ischemic index event.

#### 9.3.2 Outcomes

#### 9.3.2.1 Primary outcomes

#### Primary outcome

- Safety: SICH per SITS-MOST definition
- Mortality (mRS=6) within 90 days
- Outcome: Functional Independency as defined by mRS 0-2 within 90 days

A modified Rankin score, mRS, is used to evaluate daily activity of the patient at day 90 (described in Attachment 8.3). The scores are entered in the on-line entry form. The score 0-1 is defined as favourable outcome and 0-2 as independence of the patient.

Symptomatic intracerebral haemorrhage, SICH, is defined as 'Intracerebral haemorrhage' (parenchymatous haemorrhage type 2, PH2), at the 22-36 hours post-treatment scan combined with neurological deterioration leading to an increase of 4 points on the NIH Stroke Scale' (SITS-MOST definition).

The evaluation of post-treatment haemorrhage is done using the CT/MRI scan performed between 22-36 hours after start of treatment or earlier if clinically indicated.

Death within 90 days as classified by the investigator according to cause: cerebral infarct, cerebral haemorrhage, cerebral infarct and haemorrhage unspecified, myocardial infarct, pulmonary embolism, pneumonia, other vascular cause, unknown and other cause of death (ICD 10 to be provided).

#### 9.3.2.2 Secondary outcomes

#### Secondary outcomes

- Patient characteristics at baseline including stroke severity (NIHSS)
  - Outcomes: Favourable outcome as defined by mRS 0-1 within 90 days
  - Secondary safety: SICH per ECASS 2 within 90 days
  - Delays of management
    - o Time from onset of symptoms start of treatment
    - Time from onset of symptoms door (or as captured in the registry arrival at hospital)
    - Door needle time

**Study Number 0135-0344** 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 9.3.3 Covariates

#### Specification of data collection from the index stroke event

At baseline: Demographic data (age, sex, weight), NIHSS and pre-stroke mRS, blood pressure, laboratory values (plasma glucose, cholesterol) medical history including comorbidities and concomitant medication, results of imaging scans, time logistics

At 24 hours: NIHSS score, blood pressure, laboratory and imaging scans if performed. During hospital stay: details of concomitant medications, additional imaging scans

At 7 day or discharge if occurred earlier than 7 days: Date/time discharge, NIHSS scores, blood pressure, type of stroke and AF, medications

At 3-months follow up: mRS scale, any events including recurrent stroke (haemorrhagic or ischaemic), major extracranial haemorrhage

The analysis will include standard covariates. Standard SITS-ISTR safety parameters:

- Baseline and demographic variables available in SITS for describing patient characteristics such as but not limited to stroke severity, age, gender etc. (standard covariates)
- Symptomatic intracerebral haemorrhage (SICH): Intracerebral haemorrhage (parenchymatous haemorrhage type 2), at post-treatment scan combined with neurological deterioration leading to an increase of 4 points on the NIH Stroke Scale (SITS-MOST definition)
- Mortality: Death (mRS = 6) at day 90
- Independence / favourable outcome:

Independence for the activities of daily living at day 90. Good functional outcome is defined as a modified Rankin Scale (mRS) score of both 0-2 (independence) and 0-1 (favourable) and independency / favourable outcome at 90 days (mRS 0-2, mRS 0-1

Patient management variables

- o Time from onset to door
- o Door to needle (treatment) time
  Onset to treatment time

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.4 ONSET TO TREATMENT TIME DATA SOURCES

#### Data is collected within the SITS-ISTR registry according to their standard procedures.

SITS is an academic-driven, non-profit, international collaboration. It is an initiative by the medical profession aimed at driving excellence in acute and secondary stroke treatment, and to develop new knowledge and leading research. SITS-ISTR is an ongoing, prospective, multinational and academic driven registry for centres using thrombolysis for the treatment of acute ischaemic stroke patients. The registry contains data about alteplase treatment independent of the time since stroke onset. Information related to patient demographics, baseline characteristics, stroke severity at baseline, onset to treatment time, risk factors, drug treatment history, admission time and data on baseline and follow-up imaging scans are collected in SITS-ISTR

#### 9.5 STUDY SIZE

The sample size was not based on any formal power calculation, rather chosen pragmatically in consultation with authorities and based on numbers achievable within a 3-year period. Approximately 2000 acute ischaemic patients who were treated with IV thrombolysis within 4.5 hours within symptom onset constitute the main analysis population. Data from a minimum of 500 European patients are expected within the database during post approval phase as well as equal number during the pre-approval phase in patients > 80 years old acute ischemic stroke patients.

#### 9.6 DATA MANAGEMENT

Data in the SITS registry are entered on-line through the SITS website. SITS uses the two-factors authentication to login to the registry, i.e. first by username and password and then by a code which is sent to the user either by SMS or by e-mail. Each investigator/study nurse has a personal access code which must be kept secret and used only by the owner. All data entry from a centre can be made by each member of the local team, but once the data entry is confirmed (i.e. cannot be changed), the person who made the confirmation will be identified on the data entry form.

For the purpose of analysis, a download will be made in Excel/ CSV format which will then be transferred in the appropriate advance data analysis software such as STATISTICA/ SAS.

Data collection in this study is approved as part of the SITS-ISTR study framework by the Regional Research Ethics Committee in Stockholm, Sweden. Data analyses are performed according to SITS policy and under the responsibility of the Scientific Committee.

#### 9.7 DATA ANALYSIS

A non-interventional post-approval study on SITS-ISTR existing data of intravenous rt-PA (0.9 mg/kg) in acute ischaemic stroke patients over 80 years, according to the Summary of

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Product Characteristics (SmPC) of European countries being part of the mutual recognition procedure within the academic SITS-ISTR (International Stroke Thrombolysis Registry, ongoing since December 2002).

Descriptive statistics (absolute and relative frequencies, means, standard deviations, medians, inter quartile ranges, minimum and maximum values, 95% confidence intervals and proportions, as appropriate) for baseline and demographic characteristics for all included patients will be provided. To compare demographic and clinical baseline characteristics between pre-approval and post-approval patients over >80 years, standardized differences will be used. Multivariable analyses (exploratory) with adjustment for differences or imbalances in prognostic variables for outcome comparison will be performed.

#### 9.7.1 Main analysis

We will compare the outcome of interest both in unmatched and propensity score matched patient sets as described below. The primary analysis will be on propensity score matched patient sets and we will compare the post-approval >80 year old patients with the pre-approval retrospective >80 year olds regarding baseline demographics, clinical and radiological parameters, as well as treatment logistics, safety outcomes, functional outcome and death. Secondary analysis will be on unmatched patient sets, i.e. all patients fulfilling the inclusions-exclusions criteria will be included in this analysis. A sensitivity analysis restricted to European and non-European patients might be considered if minimum sample size required for analysis is met in the matched patient set.

Patient sets analysed includes "unmatched" and "matched". "Unmatched" patients set composed of IV thrombolysis treated patients >80 years from both pre-approval and post-approval phase those who fulfil the inclusions-exclusions criteria. Matched patient set constitute propensity score matched pair (1:1 greedy nearest neighbour matching using calipers equal to 0.2\*SD of the logit of the propensity score).

The incidence rate and corresponding 95% CI of patients with primary and secondary outcome events will be calculated within the following cohorts:

- a) Patients >80 years after approval
- b) Patients >80 years before approval

The incidence rate for the outcome of interest using as-treated approach will be calculated on the unmatched (all eligible patients) and the matched patient sets.

In the primary analysis, post-approval >80 year old patients will be matched to pre-approval >80 year old patients using a structured, iterative propensity score model with the primary objective to maximize the balance in the distribution of possible confounders between these two groups [9].

In the propensity score-matching algorithm, all baseline characteristics will be included. The corresponding propensity score of the post-approval >80 years group will be calculated for

**Study Number 0135-0344** 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

each subject and a nearest neighbour matching algorithm will then be used to match patients in the post-approval >80 years group to patients in the pre-approval >80 years group within 0.2\*SD of the logit of the propensity score. To determine whether the propensity score approach achieved balance in all potential confounders, we will compare all baseline characteristics of patients in the post-approval >80 years group to their propensity score matched pre-approval >80 year old patients using standardized difference.

We will also compare baseline characteristics between the unmatched and propensity matched subgroups to detect potential imbalances between the two populations. Differences of outcome between post-approval >80 years and pre-approval >80 years will be evaluated with univariable and multivariable binary logistic regression models adjusting for potential confounders. In these models the factors that contribute to the outcome of interest in the initial univariable analyses at p values <0.1, will be included in the multivariable model as candidate variables. The final variables that will be independently associated in the multivariable logistic regression analyses with the outcome of interest will be selected by backward stepwise selection procedures using a p value <0.05.



#### 9.8 QUALITY CONTROL

European Stroke Centres (approx. 60) continuously registering patients into SITS-ISTR having

- a typical experience from acute stroke treatment
- high quality (at least 90% complete data entered at acute phase and 70% data entered at 3m follow up) in both prospective and retrospective groups
- a willingness to participate in SITS-IVT>80 years registry

#### 9.8.1 Investigators and local procedures

According to the current processes in SITS described on the SITS web site (www.sitsinternational.org) the following persons are involved;

#### National Coordinator

A National Coordinator (NC) is appointed by SITS as to be the responsible person for the SITS activity in the specific country. The NC has an overview of the infrastructure in regards to stroke care treatments in the country. The role of NC is to coordinate among the different centers in the country. SITS has engaged leading stroke scientists as National Coordinators in each participating country.

#### Local coordinator/ Centre coordinator

The Local Coordinator (LC) is responsible for the centre activity and ultimate responsibility of the data entered in the SITS registry from the hospital. The LC must be a doctor authorised by the medical head of the department.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Local user

The Local User (LU) is responsible for entering data in the SITS registry. The LU must be appointed by the LC and operating within the stroke unit.

Internal data quality controls will be done by the SITS Coordinating Office, which will include:

- 1. Validation rules for key data parameters so that impossible data will not be possible to enter
- 2. Online monitoring to find out inconsistent data entry, data completeness
- 3. In addition to online data monitoring, inconsistency and completeness check every 6 months. Normally investigators are informed by newsletter regarding the completeness of data entry for overall registry and asked to complete the missing data. In case of major inconsistency or high rate of missing data investigators are contacted personally by e-mail.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

#### Non-interventional study based on existing data

The quality of a study based on existing data relies on accuracy of recorded data. Important data may not be available.

#### **Selection bias**

There is a risk of selection bias at the patient level. Sites might preferentially include "interesting" cases to the SITS study. To minimize selection bias at the patient level, centres were reminded by e-mail every 3 months that all consecutive patients from each site who meet entry criteria must be included in the SITS-Registry.

#### Lost to follow up

As with all observational studies a loss to follow up can occur. In this study this will affect the patients with a pre-planned follow up (patients initiating IV thrombolysis within the 3 months after the index event). However, considering the short time period of the follow up and the lost to follow up at 3 months in the general SITS Registry being 20%, a similar percentage of lost to follow up is expected in this study as well.

For the analysis of clinical outcome events we do not exclude patients lost to follow-up after IV thrombolysis initiation and before the 3 months after index event, which could lead to underidentification of clinical outcome events.

#### 9.10 OTHER ASPECTS

Not applicable.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.11 SUBJECTS

**Study Number 0135-0344** 

Patients over 80 years old presenting with acute ischaemic stroke symptoms for which thrombolysis treatment was initiated within 4.5 hours after stroke onset according to the SmPC during the study period June 2015 to June 2021 divided into pre-approval (June 2015 to June 2018) and post-approval (July 2018 to June 2021).

#### 9.11.1 Cases

Not applicable.

#### **9.11.2** Controls

Please refer to Section 9.7.1

#### 9.12 **BIAS**

To assess potential channeling bias, baseline characteristics of all patients fulfilling the in/exclusion criteria and were included in SITS-ISTR registry in the defined time period will be described based on the IV thrombolysis treatment they receive for ischemic stroke within 4.5 hours from symptoms onset.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. PROTECTION OF HUMAN SUBJECTS

Regulated under the SITS ISTR registry. All data entered into the SITS International Thrombolysis registry are encrypted in order to maintain patient data privacy. The individual patient and its research data is identified by a unique registry identification number. Access to data is strictly controlled by permitting two-way authentication, i.e. each user a unique username and password and a code received by sms or e-mail. Additionally, each user has restrictions in viewing data sets, depending on their activity role in the database. Each data entry is centrally monitored by internal quality checks, such as automatic range checks and a full audit trail is maintained.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

According to the European Medicines Agency (EMA) Guideline on Good Pharmacovigilance Practices (GVP), Adverse Event (AE) reporting is not required for Non-Interventional Study (NIS) which is based on secondary data use.

12. AS AN OBSERVATIONAL STUDY, BASED ON EXISTING DATA, ALL PATIENT DATA IS DE-IDENTIFIED AND WILL BE ANALYSED IN AGGREGATE. INDIVIDUAL PATIENT SAFETY RELATED INFORMATION WILL NOT BE CAPTURED DURING THIS STUDY. THUS, INDIVIDUAL SAFETY REPORTING IS NOT APPLICABLE. SAFETY REPORTING WILL BE DONE CUMULATIVELY IN AGGREGATE IN THE STUDY REPORT.PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The results will be disclosed on EnCEPP, Publications will be prepared and the full study report will be submitted to the authorities.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 13. REFERENCES

.

#### 13.1 PUBLISHED REFERENCES

*Include references with P, R, and S numbers here.* 

- 1. Johnson W, Onuma O, Owolabi M, Sachdev S. Stroke: a global response is needed. Bull World Health Organ. Switzerland2016. p. 634-a.
- 2. Feigin VL et al. Atlas of the global burden of stroke (1990-2013): The GBD 2013 Study. Neuroepidemiology 2015; 45(3):230-6
- 3. Wahlgren NG. Introduction to Karolinska Stroke Update 2000. In: Update on Stroke Therapy 2000-2001, NG Wahlgren, ed, Karolinska Stroke Update, Stockholm, 2001; 17-19.
- 4. Menken M, Munsat TL, Toole JF. The global burden of disease study. Implications for neurology. Arch Neurol. 2000; 57: 418–420.
- 5. Indredavik B, Bakke F, Slordahl SA, Rokseth R, Haheim LL. Stroke unit treatment. 10-year follow up. Stroke 1999; 8;1524-7
- 6. Chan DKY, Cordato D, O'Rourke F, Chan DL, Pollack M, Middleton S, et al. Comprehensive stroke units: A review of comparative evidence and experience. International Journal of Stroke. 2013;8:260-264
- 7. The National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group: Tissue plasminogen activator for acute ischemic stroke. New Engl J Med 1995;333:1581-1587.
- 8. Hacke W, Donnan G, Fieschi C, Kaste M, von Kummer R, Broderick JP, Brott T, Frankel M, Grotta JC, Haley EC Jr, Kwiatkowski T, Levine SR, Lewandowski C, Lu M,Lyden P, Marler JR, Patel S, Tilley BC, Albers G: Association of outcome with early stroke treatment: pooled analysis of ATLANTIS, ECASS, and NINDS rt-PA stroke trials. Lancet 2004;363:768-774
- 9. Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, et al. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a metaanalysis of individual patient data from randomised trials. Lancet. 2014;384(9958):1929-35
- 10. Wahlgren N, Ahmed N, Davalos A, Ford GA, Grond M, Hacke W, Hennerici MG, Kaste M, Kulkens S, Larrue V, Lees KR, Roine RO, Soinne L, Toni D, Vanhooren G: Thrombolysis with alteplase for acute ischaemic stroke in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST): an observational study. Lancet 2007;369:275-282.
- 11. Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D, for the ECASS Investigators. Thrombolysis with Alteplase 3 to 4.5 Hours after Acute Ischemic Stroke. New Engl J Med 2008; 359: 1317-1329.

- 12. Wahlgren N, Ahmed N, Davalos A, Hacke W, Millan M, Muir K, Roine RO, Toni D, Lees KR. Thrombolysis with alteplase 3-4.5 h after acute ischaemic stroke (SITS-ISTR): an observational study. Lancet 2008; 372: 1303-1309.
- 13. Berkhemer OA, Fransen PS, Beumer D et al. A randomized trial of intraarterial treatment for acute ischaemic stroke. N Engl J Med 2015; 372: 11–20.
- 14. Goyal M, Demchuk AM, Menon BK et al. Randomized assessment of rapid endovascular treatment of ischaemic stroke. N Engl J Med 2015; 372: 1019–30.
- 15. Campbell BC, Mitchell PJ, Kleinig TJ et al. Endovascular therapy for ischaemic stroke with perfusion-imaging selection. N Engl J Med 2015; 372: 1009–18.
- 16. Saver JL, Goyal M, Bonaf\_e A et al. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med 2015; 372: 2285–95.
- 17. Jovin TG, Chamorro \_A, Cobo E et al. Thrombectomy within 8 hours after symptom onset in Ischaemic stroke. N Engl J Med 2015; 372: 2296–306.
- 18. Wahlgren N, Moreira T, Michel P, et al; for ESO-KSU, ESO, ESMINT, ESNR and EAN. Mechanical thrombectomy in acute ischemic stroke: Consensus statement by ESO-Karolinska Stroke Update 2014/2015, supported by ESO, ESMINT, ESNR and EAN. Int J Stroke. 2016 Jan;11(1):134-47.
- 19. Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Dávalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, ereira VM, Rempel J, Millán M, Davis SM, Roy D, Thornton J, Román LS, Ribó M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators.. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. PubMed PMID: 26898852.
- 20. Socialstyrelsen. Nationella riktlinjer för strokesjukvård 2009 stöd för styrning och ledning. 2009.
- 21. Powers WJ, Derdeyn CP, Biller J, Coffey CS, Hoh BL, Jauch EC, et al. 2015 american heart association/american stroke association focused update of the 2013 guidelines for the early management of patients with acute ischemic stroke regarding endovascular treatment: A guideline for healthcare professionals from the american heart association/american stroke association. Stroke. 2015;46:3020-3035
- 22. Hossman KA. Pathophysiology of cerebral infarction. In: Wilken PJ, Bruyn GW, Klawans HL, eds. Handbook of Clinical Neurology, Vol 53. Amsterdam, Elsevier Science Publishers 1988, 107-153
- 23. Hacke W, Kaste M, Fieschi C, et al, and the European Cooperative Acute Stroke Study (ECASS). Intravenous thrombolysis with recombinant tissue plasminogen activator for acute hemispheric stroke. JAMA 1995; 274: 1017–25.
- 24. Hacke W, Kaste M, Fieschi C, et al. Randomised double-blind placebo-controlled trial of thrombolytic therapy with intravenous alteplase in acute ischaemic stroke (ECASS II). Lancet 1998; 352: 1245–51.

- 25. Clark WM, Wissman S, Albers GW, Jhamandas JH, Madden KP, Hamilton S, for the ATLANTIS Study Investigators. Recombinant tissue-type plasminogen activator (alteplase) for ischemic stroke 3 to 5 hours after symptom onset. The ATLANTIS Study: a randomized controlled trial. JAMA 1999; 282: 2019–26.
- 26. Davis SM, Donnan GA, Parsons MW, et al, and the EPITHET investigators. Effects of alteplase beyond 3 h after stroke in the Echoplanar Imaging Thrombolytic Evaluation Trial (EPITHET): a placebo-controlled randomised trial. Lancet Neurol 2008; 7: 299–309.
- 27. Sandercock P, Wardlaw JM, Lindley RI, et al, and the IST-3 collaborative group. The benefits and harms of intravenous thrombolysis with recombinant tissue plasminogen activator within 6 h of acute ischaemic stroke (the third international stroke trial [IST-3]): a randomised controlled trial. Lancet 2012; 379: 2352–63.
- 28. Lees KR, Bluhmki E, von Kummer R, Brott TG, Toni D, Grotta JC, Albers GW, Kaste M, Marler JR, Hamilton SA, Tilley BC, Davis SM, Donnan GA, Hacke W; ECASS, ATLANTIS, NINDS and EPITHET rt-PA Study Group, Allen K, Mau J, Meier D, del Zoppo G, De Silva DA, Butcher KS, Parsons MW, Barber PA, Levi C, Bladin C, Byrnes G. Time to treatment with intravenous alteplase and outcome in stroke: an updated pooled analysis of ECASS, ATLANTIS, NINDS, and EPITHET trials. Lancet 2010; 375:1695-703
- 29. Chiu D, Krieger D, Villar-Cordova C, Kasner SE, Morgenstern LB, Bratina PL, Yatsu FM, Grotta JC. Intravenous tissue plasminogen activator for acute ischemic stroke. Feasibility, Safety and efficacy in the first year of clinical practice. Stroke. 1998;29:18-22
- 30. Trouillas P, Nighoghossian N, Derex L, Adeleine P, Honnorat J, Neuschwander P, Riche G, Getenet JC, Li W, Froment JC, Turjman F, Malicier D, Fournier G, Gabry AL, Ledoux X, Berthezène Y, Ffrench P, Dechavanne M. Thrombolysis with intravenous rtPA in a series of 100 cases of acute carotid territory stroke. Determination of etiological, topographic, and radiological outcome factors. Stroke 1998;29:2529-40
- 31. Katzan IL, Furlan AJ, Lloyd LE, Frank JI, Harper DL, Hinchey JA, Hammel JP, Qu A, Sila CA. Use of tissue-type plasminogen activator for acute ischemic stroke. The Cleveland experience. JAMA 2000;283:1151-58
- 32. Schmülling S, Grond M, Rudolf J, Heiss WD. One-year follow-up in acute stroke patients treated with rtPA in clinical routine. Stroke 2000;31:1552-54
- 33. Albers GW, Bates VE, Clark WM, Bell R, Verro P, Hamilton SA. Intravenous tissuetype plasminogen activator for treatment of acute stroke. The standard treatment with alteplase to reverse stroke (STARS) study. JAMA 2000;283:1145-50
- 34. Tanne D, Demchuk A., Kasner SE, Grond M, Hanson S, Hamilton S, Buchan AM, Wang DZ, Wechsler LR, Zweifler R, Levine SR, for the t-PA in acute stroke collaborators. A large multinational investigation to predict t-PA related symptomatic ICH in patients with acute ischemic stroke. Stroke 30, 248, 1999

- 35. Ford GA, Ahmed N, Azevedo E, et al. Intravenous alteplase for stroke in those older than 80 years old. Stroke. 2010 Nov;41(11):2568-74. doi: 10.1161/STROKEAHA.110.581884. Epub 2010 Oct 7. PubMed PMID: 20930163.
- 36. Mishra NK, Ahmed N, Andersen G, et al; VISTA collaborators; SITS collaborators. Thrombolysis in very elderly people: controlled comparison of SITS International Stroke Thrombolysis Registry and Virtual International Stroke Trials Archive. BMJ. 2010 Nov 23;341:c6046. doi: 10.1136/bmj.c6046.. PubMed PMID: 21098614; PubMed Central PMCID: PMC2990864.
- 37. Whiteley WN, Emberson J, Lees KR, et al; Stroke Thrombolysis Trialists' Collaboration.. Risk of intracerebral hemorrhage with alteplase after acute ischaemic stroke: a secondary analysis of an individual patient data meta-analysis. Lancet Neurol. 2016 Aug;15(9):925-33. doi: 10.1016/S1474-4422(16)30076-X.
- 38. ESO Guidelines: webpage: eso-stroke.org/eso-stroke/education/education-guidelines.html, ESO guideline Updated 2009)
- 39. Demaerschalk BM, Kleindorfer DO, Adeoye OM, et al; American Heart Association Stroke Council and Council on Epidemiology and Prevention. Scientific Rationale for the Inclusion and Exclusion Criteria for Intravenous Alteplase in Acute Ischemic Stroke: A Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Feb;47(2):581-641. doi: 10.1161/STR.000000000000086. Epub 2015 Dec 22. Review. PubMed PMID: 26696642
- 40. Ahmed N, Lees KR, Ringleb PA, Bladin C, Collas D, Toni D, Ford GA; The SITS Investigators. Outcome after stroke thrombolysis in patients >80 years treated within 3 hours vs >3-4.5 hours. Neurology. 2017 Oct 10;89(15):1561-1568. doi:10.1212/WNL.0000000000004499. Epub 2017 Sep 8. PubMed PMID: 28887377

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>Reference Number | Date | Title |
|---|---|---|---|
| 1 | not applicable | September 2019 | common-<br>combined-Actilyse-<br>en-clean-September<br>2019 |
| 2 | not applicable | September 2019 | SITS- IVTP<br>Standard data entry<br>form_2019<br>September |
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# ANNEX 2. ENCEPP CECKLIST FOR STUDY PROTOCOLS

A copy of the ENCePP Checklist for Study protocols available at website: encepp.eu/standards and guidances/index.html completed and signed by the main author of

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



Doc.Ref. EMA/540136/2009



# **ENCePP Checklist for Study Protocols (Revision 4)**

Adopted by the ENCePP Steering Group on 15/10/2018

The European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) welcomes innovative designs and new methods of research. This Checklist has been developed by ENCEPP to stimulate consideration of important principles when designing and writing a pharmacoepidemiological or pharmacovigilance study protocol. The Checklist is intended to promote the quality of such studies, not their uniformity. The user is also referred to the ENCePP Guide on Standards in Pharmacoepidemiology, which reviews and gives direct electronic access to guidance for research in pharmacoepidemiology and pharmacovigilance.

For each question of the Checklist, the investigator should indicate whether or not it has been addressed in the study protocol. If the answer is "Yes", the section number of the protocol where this issue has been discussed should be specified. It is possible that some questions do not apply to a particular study (for example, in the case of an innovative study design). In this case, the answer 'N/A' (Not Applicable) can be checked and the "Comments" field included for each section should be used to explain why. The "Comments" field can also be used to elaborate on a "No" answer.

This Checklist should be included as an Annex by marketing authorisation holders when submitting the protocol of a non-interventional post-authorisation safety study (PASS) to a regulatory authority (see on the format and content of the protocol of non-interventional udies). The Checklist is a supporting document and does not replace the format of the protocol for PASS presented in the Guidance and Module VIII of the Good pharmacovigilance practices (GVP).

#### Study title:

Safe Implementation of Treatments in Stroke (SITS) -

Intravenous thrombolysis in acute ischaemic stroke patients over 80 years, SITS-IVT>80 years study

| EU PAS Register® number: |
|---------------------------------------------|
| Study reference number (if applicable): n/a |

| Sect | tion 1: Milestones | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 1.1 | Does the protocol specify timelines for | | | | |
| | 1.1.1 Start of data collection <sup>1</sup> | $\boxtimes$ | | | 6 |
| | 1.1.2 End of data collection <sup>2</sup> | | | | 6 |
| | 1.1.3 Progress report(s) | | | | |
| | 1.1.4 Interim report(s) | | | | 6 |
| | 1.1.5 Registration in the EU PAS Register® | | | | 6 |

<sup>1</sup> Date from which information on the first study is first recorded in the study dataset or, in the case of secondary use of data, the date from which data extraction starts.

<sup>2</sup> Date from which the analytical dataset is completely available.



Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Sec | tion 1: Milestones | Yes | No | N/A | Section |
|---|---|---|---|---|---|
| | 1.1.6 Final report of study results. | | | | 6 |
| Соп | nments: | | | | |
| Sec | tion 2: Research question | Yes | No | N/A | Section |
| 2.1 | Does the formulation of the research question and objectives clearly explain: | | | | 8 |
| | 2.1.1 Why the study is conducted? (e.g. to address an important public health concern, a risk identified in the risk management plan, an emerging safety issue) | | | | 8 |
| | 2.1.2 The objective(s) of the study? | | | | 8 |
| | 2.1.3 The target population? (i.e. population or subgroup to whom the study results are intended to be generalised) | | | | 8 |
| | 2.1.4 Which hypothesis(-es) is (are) to be tested? | | | | 8 |
| | 2.1.5 If applicable, that there is no a priori<br>hypothesis? | | | | |
| Com | ments: | | | | |
| Sec | tion 3: Study design | Yes | No | N/A | Section<br>Number |
| 3.1 | Is the study design described? (e.g. cohort, case-<br>control, cross-sectional, other design) | $\boxtimes$ | | | 9.1 |
| 3.2 | Does the protocol specify whether the study is<br>based on primary, secondary or combined data<br>collection? | | | | 9.1 |
| 3.3 | Does the protocol specify measures of occurrence? (e.g., rate, risk, prevalence) | | | | 9.3 |
| 3.4 | Does the protocol specify measure(s) of association? (e.g. risk, odds ratio, excess risk, rate ratio, hazard ratio, risk/rate difference, number needed to harm (NNH)) | | | | 9.3 |
| 3.5 | Does the protocol describe the approach for the collection and reporting of adverse events/adverse reactions? (e.g. adverse events that will not be collected in case of primary data collection) | | | | 11 |
| Com | ments: | | | | |
| Cool | ion 4: Source and study populations | Yes | No | N/<br>A | Section<br>Number |
| | | $\boxtimes$ | | | 9.2 |
| 4.1 | Is the source population described? | | | | |
| 4.1<br>4.2 | Is the planned study population defined in terms of: | 1 | | | |
| 4.1 | Is the planned study population defined in terms | | | | 9.1<br>9.1 |

ENCePP Checklist for Study Protocols (Revision 4)

Page 2/6



Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Sec | tion 4: Source and study populations | Yes | No | N/<br>A | Section |
|---|---|---|---|---|---|
| | 4.2.3 Country of origin | | | | 9.1 |
| | 4.2.4 Disease/indication | | | | 9.1 |
| | 4.2.5 Duration of follow-up | $\boxtimes$ | | | 9.1 |
| 4.3 | Does the protocol define how the study population will be sampled from the source population? (e.g. event or inclusion/exclusion criteria) | | | | 9 |
| Con | nments; | | | | |
| Sec | tion 5: Exposure definition and measurement | Yes | No | N/A | Section |
| 5.1 | Does the protocol describe how the study exposure is defined and measured? (e.g. operational details for defining and categorising exposure, measurement of dose and duration of drug exposure) | × | | | 9.1 |
| 5.2 | Does the protocol address the validity of the exposure measurement? (e.g. precision, accuracy, use of validation sub-study) | × | | | 7 |
| 5.3 | Is exposure categorised according to time windows? | | | | 9.2 |
| 5.4 | Is intensity of exposure addressed?<br>(e.g. dose, duration) | | | | 7 |
| 5.5 | Is exposure categorised based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | | | 7 |
| 5.6 | Is (are) (an) appropriate comparator(s) identified? | | | | |
| | tion 6: Outcome definition and measurement | Van | No | 21/2 | C |
| 3CC | tion o. Outcome definition and measurement | Yes | No | N/A | Section<br>Number |
| 6.1 | Does the protocol specify the primary and<br>secondary (if applicable) outcome(s) to be<br>investigated? | | | | 9.2 |
| 6.2 | Does the protocol describe how the outcomes are defined and measured? | | | | 9.3 |
| 6.3 | Does the protocol address the validity of outcome<br>measurement? (e.g. precision, accuracy, sensitivity,<br>specificity, positive predictive value, use of validation sub-<br>study) | | | | 9.3 |
| 6.4 | Does the protocol describe specific outcomes relevant for Health Technology Assessment? (e.g. HRQoL, QALYs, DALYS, health care services utilisation, burden of disease or treatment, compliance, disease management) | | | | |
| Com | ments: | | | | |

H

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Sec | tion 7: Bias | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 7.1 | Does the protocol address ways to measure confounding? (e.g. confounding by indication) | | | | 9.7 |
| 7.2 | Does the protocol address selection bias? (e.g. healthy user/adherer bias) | | | | 9.9 |
| 7.3 | Does the protocol address information bias?<br>(e.g. misclassification of exposure and outcomes, time-related<br>bias) | | | | |
| Com | ments: | | | | |
| Sec | tion 8: Effect measure modification | Yes | No | N/A | Section |
| | The state of the s | 163 | 140 | III/A | Number |
| 8.1 | Does the protocol address effect modifiers?<br>(e.g. collection of data on known effect modifiers, sub-group<br>analyses, anticipated direction of effect) | | | | |
| Com | ments: | | | | |
| Sec | tion 9: Data sources | Yes | No | N/A | Section |
| | | | | | Number |
| 9.1 | Does the protocol describe the data source(s) used<br>in the study for the ascertainment of: | | | | |
| | 9.1.1 Exposure? (e.g. pharmacy dispensing, general<br>practice prescribing, claims data, self-report, face-to-face<br>interview) | | | | 9.6 and 9.8 |
| | 9.1.2 Outcomes? (e.g. clinical records, laboratory markers<br>or values, claims data, self-report, patient interview<br>including scales and questionnaires, vital statistics) | | | | 9.6 and 9.8 |
| | 9.1.3 Covariates and other characteristics? | | | | 9.6 and 9.8 |
| 9.2 | Does the protocol describe the information available from the data source(s) on: | | | | |
| | <ol> <li>Exposure? (e.g. date of dispensing, drug quantity,<br/>dose, number of days of supply prescription, daily dosage,<br/>prescriber)</li> </ol> | ⊠ | | | |
| | 9.2.2 Outcomes? (e.g. date of occurrence, multiple event, severity measures related to event) | $\boxtimes$ | | | |
| | <ol> <li>9.2.3 Covariates and other characteristics? (e.g. age,<br/>sex, clinical and drug use history, co-morbidity, co-<br/>medications, lifestyle)</li> </ol> | | | | |
| 9.3 | Is a coding system described for: | | | | |
| | 9.3.1 Exposure? (e.g. WHO Drug Dictionary, Anatomical<br>Therapeutic Chemical (ATC) Classification System) | | | ⊠ | |
| | <ol> <li>9.3.2 Outcomes? (e.g. International Classification of<br/>Diseases (ICD), Medical Dictionary for Regulatory Activities<br/>(MedDRA))</li> </ol> | | | ⋈ | |
| | 9.3.3 Covariates and other characteristics? | | | | |
| | Is a linkage method between data sources | 1000 | | | |

ENCePP Checklist for Study Protocols (Revision 4)

Page 4/6

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Numl 10.1 Are the statistical methods and the reason for their choice described? 10.2 Is study size and/or statistical precision estimated? 10.3 Are descriptive analyses included? 10.4 Are stratified analyses included? 10.5 Does the plan describe methods for analytic control of confounding? 10.6 Does the plan describe methods for analytic control of outcome misclassification? 10.7 Does the plan describe methods for handling missing data? 10.8 Are relevant sensitivity analyses described? 10.9 Are relevant sensitivity analyses described? 11.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? 12.3 Does the protocol discuss study feasibility? 12.4 Does the protocol discuss study feasibility? 12.5 Does the protocol discuss study feasibility? 12.6 Activity size anticipated decrease and the displayed of such sizes, validation sub-study, use of validation and external data, analytical methods). | | | | | | |
|---|---|---|---|---|---|---|
| choice described? 10.2 Is study size and/or statistical precision estimated? 10.3 Are descriptive analyses included? 10.4 Are stratified analyses included? 10.5 Does the plan describe methods for analytic control of confounding? 10.6 Does the plan describe methods for analytic control of outcome misclassification? 10.7 Does the plan describe methods for handling missing data? 10.8 Are relevant sensitivity analyses described? 10.9 Are relevant sensitivity analyses described? 10.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.1 Does the protocol from the study results? 11.3 Is there a system in place for independent review of study results? 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.1 Does the protocol discuss study feasibility? (e.g. study size, anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | Sect | tion 10: Analysis plan | Yes | No | N/A | Section |
| 10.3 Are descriptive analyses included? 10.4 Are stratified analyses included? 10.5 Does the plan describe methods for analytic control of confounding? 10.6 Does the plan describe methods for analytic control of outcome misclassification? 10.7 Does the plan describe methods for handling missing data? 10.8 Are relevant sensitivity analyses described? 10.9 No N/A Section 11: Data management and quality control with missing data? 10.9 No N/A Section 11: Data management and quality control with missing data? 10.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.1 Does the protocol growide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.1 Does the protocol discuss study feasibility? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). | 10.1 | | ⊠ | | | 9.7 |
| 10.4 Are stratified analyses included? 10.5 Does the plan describe methods for analytic control of confounding? 10.6 Does the plan describe methods for analytic control of outcome misclassification? 10.7 Does the plan describe methods for handling missing data? 10.8 Are relevant sensitivity analyses described? 10.9 No N/A Section 11: Data management and quality control of outcome misclassification? 10.9 No N/A Section 11: Data management and quality control of outcome misclassification? 10.8 Are relevant sensitivity analyses described? 10.9 No N/A Section 11: Data management and quality control of outcoments: 11.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). | 10.2 | Is study size and/or statistical precision estimated? | | | | 9.5 |
| 10.5 Does the plan describe methods for analytic control of confounding? 10.6 Does the plan describe methods for analytic control of outcome misclassification? 10.7 Does the plan describe methods for handling missing data? 10.8 Are relevant sensitivity analyses described? 10.8 Are relevant sensitivity analyses described? 10.9 No N/A Section 11: Data management and quality control Yes No N/A Section 12: Limitations Yes No N/A Section 13: Limitations 11.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Selection bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | 10.3 | Are descriptive analyses included? | | | | 9.7 |
| 10.6 Does the plan describe methods for analytic control of outcome misclassification? 10.7 Does the plan describe methods for handling missing data? 10.8 Are relevant sensitivity analyses described? 10.8 Are relevant sensitivity analyses described? 10.9 No N/A Section 11: Data management and quality control Yes No N/A Section 11: Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 12.1 Section 12: Limitations 13. Is there a system in place for independent review of study results? 14. I Does the protocol discuss the impact on the study results of: 15. 12. I Does the protocol discuss the impact on the study results of: 16. 12. I Does the protocol discuss the impact on the study results of: 17. 18. Residual/unmeasured confounding? 18. 19. 9. 9 | 10.4 | Are stratified analyses included? | | | | 9.7 |
| of outcome misclassification? 10.7 Does the plan describe methods for handling missing data? 10.8 Are relevant sensitivity analyses described? Comments: Section 11: Data management and quality control with the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? Comments: Section 12: Limitations Yes No N/A Section | 10.5 | | | | | 9.7 |
| missing data? 10.8 Are relevant sensitivity analyses described? | 10.6 | | ⊠ | | | 9.8 |
| Section 11: Data management and quality control 11.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? Comments: Section 12: Limitations Section 12: Limitations Yes No N/A Section N/A Se | 10.7 | | | | | 9.8 |
| Section 11: Data management and quality control 11.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? Comments: Section 12: Limitations Section 12: Limitations Yes No N/A Section 12: Limitations Yes No N/A Section 12: Limitations Yes No N/A Section 12: Limitations Yes No N/A Section 12: Limitations 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | 10.8 | Are relevant sensitivity analyses described? | | | | 9.7 |
| storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? Comments: Section 12: Limitations 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | Sect | ion 11: Data management and quality control | Yes | No | N/A | Section |
| 11.2 Are methods of quality assurance described? 11.3 Is there a system in place for independent review of study results? Comments: Yes No N/A Section | 11.1 | storage? (e.g. software and IT environment, database | | | | 9.2 |
| 11.3 Is there a system in place for independent review of study results? Comments: Yes No N/A Section 12: Limitations | 11.2 | | Ø | | | 9.8 |
| Section 12: Limitations 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | 11.3 | | | | | 3 |
| Number 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | Com | ments: | | | | |
| 12.1 Does the protocol discuss the impact on the study results of: 12.1.1 Selection bias? 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | Sect | ion 12: Limitations | Yes | No | N/A | Section |
| 12.1.2 Information bias? 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | 12.1 | | | | | Trumb Cr |
| 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) 9.7 | | 12.1.1 Selection bias? | | | | 9.9 |
| (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). 2.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) 9.7 | | | $\boxtimes$ | | | 9.9 |
| (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) 9.5 | | (e.g. anticipated direction and magnitude of such biases,<br>validation sub-study, use of validation and external data, | | | | 9.7 |
| comments: | 2.2 | (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the | | | × | 9.5 |
| orininents: | comi | ments: | | | | |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Sect | tion 10: Analysis plan | Yes | No | N/A | Section |
|---|---|---|---|---|---|
| 10.1 | Are the statistical methods and the reason for their choice described? | ⊠ | | | 9.7 |
| 10.2 | Is study size and/or statistical precision estimated? | | | | 9.5 |
| 10.3 | Are descriptive analyses included? | $\boxtimes$ | | | 9.7 |
| 10.4 | Are stratified analyses included? | | | | 9.7 |
| 10.5 | Does the plan describe methods for analytic control of confounding? | | | | 9.7 |
| 10.6 | Does the plan describe methods for analytic control of outcome misclassification? | | | | 9.8 |
| 10.7 | Does the plan describe methods for handling missing data? | | | | 9.8 |
| 10.8 | Are relevant sensitivity analyses described? | | | | 9.7 |
| | Does the protocol provide information on data | Yes | No | N/A | Section<br>Number |
| 11.1 | Does the protocol provide information on data<br>storage? (e.g. software and IT environment, database | | | | 9.2 |
| | maintenance and anti-fraud protection, archiving) | 573 | | | |
| | Are methods of quality assurance described? | | | | 9.8 |
| 11.5 | Is there a system in place for independent review<br>of study results? | | | | 3 |
| Com | ments: | | | | |
| Sect | ion 12: Limitations | Yes | No | N/A | Section<br>Number |
| 12.1 | Does the protocol discuss the impact on the study results of: | | | | |
| | 12.1.1 Selection bias? | $\boxtimes$ | | | 9.9 |
| | 12.1.2 Information bias? | $\boxtimes$ | | | 9.9 |
| | 12.1.3 Residual/unmeasured confounding?<br>(e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). | ⊠ | | | 9.7 |
| 2.2 | Does the protocol discuss study feasibility?<br>(e.g. study size, anticipated exposure uptake, duration of<br>follow-up in a cohort study, patient recruitment, precision of the<br>estimates) | | | × | 9.5 |
| comr | ments: | | | | |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 3. ADDITIONAL INFORMATION

#### National Institute of Health Stroke Scale, NIHSS

The NIH stroke scale, NIHSS, is described in Attachment 1.1. The scores are entered in the on-line entry form.

#### Global Evaluation Scale, GES

The Global Outcome Evaluation Scale, is described in Attachment 1.2 and the questions to answer are specified at the on-line entry form.

### **Modified Rankin Scale (Mrs)**

mRS is described in Attachment 1.3 and the questions to answer are specified at the on-line entry form

#### Brain CT/MR scan

All CT/MR scans are reviewed at the participating centre according to the local routine procedure and the outcome of the evaluation is entered in the database.

# • Baseline readings

The CTs will be evaluated with respect to haemorrhage, any sign of acute cerebral ischemic injury in the symptomatic vascular territory, or other pathology. Preferably, CTA (CT angiography) imaging will be used for identification of cerebral artery occlusion.

• Day 2 readings (22-36 hours after start of treatment)
Intracerebral haemorrhage, ICH, will be classified according to the SITS-ISTR data collection format.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | 0 | Alert | |
|---|---|---|---|
| 1a.Level of consciousness | 1 | Not alert, but arousable with minimal stimulation | |
| 1a.Level of consciousness | 2 | Not alert, requires repeated stimulation to attend | |
| | 3 | Coma | |
| 1b. Aslamation the month and | 0 | Answers both correctly | |
| <b>1b</b> . Ask patient the month and | 1 | Answers one correctly | |
| their age | 2 | Both incorrect | |
| 1 - A -1 | 0 | Obeys both correctly | |
| <b>1c</b> .Ask patient to open/close eyes and form/release fist | 1 | Obeyrs one correctly | |
| eyes and form/release list | 2 | Both incorrect | |
| 2 D | 0 | Normal | |
| 2.Best gaze (only horisontal | 1 | Partial gaze palsy | |
| eye movements) | 2 | Forced gaze deviation | |
| | 0 | No visual field loss | |
| 2.37' 1.0' 114 4' | 1 | Partial hemianopia | |
| <b>3.</b> Visual field testing | 2 | Complete hemianopia | |
| | 3 | Bilateral hemianopia (blind, incl. Cortical blindness) | |
| | 0 | Normal symmetrical movement | |
| 4. Facial paresis (Ask patient | 1 | Minor paralysis (flattened nasolabial fold, asymmetry on smiling), | |
| to show teeth or raise | 2 | Partial paralysis (total or near total paralysis of lower face) | |
| eyebrows and close eyes | _ | Complete paralysis of one or both sides (abscence of facial movement in the | |
| tightly) | 3 | upper and lower face) | |
| | 0 | Normal (extends arm 90 or 45 for 10 sec without drift) | 1 |
| | 1 | Drift | 1 |
| <b>5a.</b> Motor function | 2 | Some effort against gravity | |
| - right arm | 3 | No effort against gravity | |
| | 4 | No movement | |
| | 9 | Untestable (joint fused or limb amputated) | |
| | 0 | Normal (extends arm 90 or 45 for 10 sec without drift) | |
| | 1 | Drift | |
| <b>5b.</b> Motor Function | 2 | Some effort against gravity | |
| - left arm | 3 | No effort against gravity | |
| | 4 | No movement | |
| | 9 | Untestable (joint fused or limb amputated) | |
| | 0 | Normal (holds leg in 30 position for 5 sec without drift) | |
| | 1 | Drift | |
| <b>6a.</b> Motor Function - right leg | 2 | Some effort against gravity | |
| va. Motor runction - right leg | 3 | No effort against gravity | |
| | 4 | No movement | |
| | 9 | Untestable (joint fused or limb amputated) | |
| | 0 | Normal (holds leg in 30 position for 5 sec without drift) | |
| | 1 | Drift | |
| <b>6b</b> . Motor Function – left leg | 2 | Some effort against gravity | |
| ob. Motor Function – left leg | 3 | No effort against gravity | <del> </del> |
| | 4 | No movement | - |
| | 9 | Untestable (joint fused or limb amputated) | - |
| | 0 | No ataxia | - |
| 7. Limb ataxia | | Present in one limb | - |
| 7. LIIIIO ataxia | 1 | Present in one limb Present in two limbs | - |
| Q Cangamy (van ming vi-1-4-4-4-4-4-4-4-4-4-4-4-4-4-4-4-4-4-4- | 0 | Normal | - |
| <b>8</b> . Sensory (use pinprick to test | 1 | Mild to moderate decrease in sensation | - |
| arma loca trunk and face | | iving to moderate decrease in sensation | |
| arms, legs trunk and face, | | | |
| arms, legs trunk and face, compare side to side) | 2 | Severe to total sensory loss | |
| | 2 | · | |
| compare side to side) | 2 | No aphasia | |
| 9. Best language (describe | 2<br>0<br>1 | No aphasia Mild to moderate aphasia | |
| compare side to side) | 2<br>0<br>1<br>2 | No aphasia Mild to moderate aphasia Severe aphasia | |
| 9. Best language (describe | 2<br>0<br>1<br>2<br>3 | No aphasia Mild to moderate aphasia Severe aphasia Mute | |
| 9. Best language (describe picture, name items) | 2<br>0<br>1<br>2<br>3<br>0 | No aphasia Mild to moderate aphasia Severe aphasia Mute Normal articulation | |
| 9. Best language (describe picture, name items) 10. Dysarthria (read several | 2<br>0<br>1<br>2<br>3<br>0<br>1 | No aphasia Mild to moderate aphasia Severe aphasia Mute Normal articulation Mild to moderate slurring of words | |
| 9. Best language (describe picture, name items) | 2<br>0<br>1<br>2<br>3<br>0<br>1<br>2 | No aphasia Mild to moderate aphasia Severe aphasia Mute Normal articulation Mild to moderate slurring of words Near unintelligible or unable to speak | |
| 9. Best language (describe picture, name items) 10. Dysarthria (read several | 2<br>0<br>1<br>2<br>3<br>0<br>1<br>2<br>9 | No aphasia Mild to moderate aphasia Severe aphasia Mute Normal articulation Mild to moderate slurring of words Near unintelligible or unable to speak Intubated or other physical barrier | |
| 9. Best language (describe picture, name items) 10. Dysarthria (read several | 2<br>0<br>1<br>2<br>3<br>0<br>1<br>2<br>9 | No aphasia Mild to moderate aphasia Severe aphasia Mute Normal articulation Mild to moderate slurring of words Near unintelligible or unable to speak Intubated or other physical barrier Normal | |
| 9. Best language (describe picture, name items) 10. Dysarthria (read several words) | 2<br>0<br>1<br>2<br>3<br>0<br>1<br>2<br>9 | No aphasia Mild to moderate aphasia Severe aphasia Mute Normal articulation Mild to moderate slurring of words Near unintelligible or unable to speak Intubated or other physical barrier Normal Inattention or extinction to bilateral simultaneous stimulation in one of the | |
| 9. Best language (describe picture, name items) 10. Dysarthria (read several words) 11. Extinction and inattention | 2<br>0<br>1<br>2<br>3<br>0<br>1<br>2<br>9 | No aphasia Mild to moderate aphasia Severe aphasia Mute Normal articulation Mild to moderate slurring of words Near unintelligible or unable to speak Intubated or other physical barrier Normal | |

**Study Number 0135-0344** 

c30353958-01

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1.2 Global evaluation scale, GES

Has a change in the patient's clinical condition occurred after treatment?

# Check one alternative:

| Much better | +2 |
|-------------|----|
| Better | +1 |
| Unchanged | 0 |
| Worse | -1 |
| Much worse | -2 |
| Dead | -3 |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1.3 Modified Rankin Scale, mRS

| Score | Description |
|---|---|
| 0 | No symptoms at all |
| 1 | No significant disability despite symptoms; able to carry out all usual duties and activities |
| 2 | Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance |
| 3 | Moderate disability; requiring some help, but able to walk without assistance |
| 4 | Moderately severe disability; unable to walk without assistance and unable to attend own bodily needs without assistance |
| 5 | Severe disability; bedridden, incontinent and requiring constant<br>nursing care and attention |
| 6 | Dead |
| Total (0-6): | |



#### APPROVAL / SIGNATURE PAGE

Document Number: c30353958 Technical Version Number: 1.0

**Document Name:** ctp-safe-implementation-of-treatments-in-stroke-sits

**Title:** CTP-Safe Implementation of Treatments in Stroke (SITS) - Intravenous thrombolysis in acute ischaemic stroke patients over 80 years, SITS-IVT>80 years study

# **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval- Established Core Products | | 25 Nov 2019 12:15 CET |
| Approval-Safety Evaluation Therapeutic Area | | 25 Nov 2019 12:24 CET |
| Approval-Team Member Medical<br>Affairs | | 25 Nov 2019 13:35 CET |
| Approval-EU Qualified Person<br>Pharmacovigilance | | 25 Nov 2019 13:41 CET |
| Approval-Pharmacovigilance | | 25 Nov 2019 14:17 CET |
| Approval-On behalf of or | | 25 Nov 2019 15:12 CET |

Boehringer IngelheimPage 2 of 2Document Number: c30353958Technical Version Number: 1.0

(Continued) Signatures (obtained electronically)

| Meaning of Signature |
|----------------------|
|----------------------|